CLINICAL TRIAL: NCT04097808
Title: Impact of the Source and Polyphenol-containing Food Matrices on the Bioavailability of Peptan® (Collagen Peptides) in Healthy Subjects
Brief Title: Impact of the Source and Food Matrices on the Bioavailability of Peptan® (Collagen Peptides) in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BTS1362/19
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-09

CONDITIONS: Bioavailability
Keywords: bioavailability; collagen peptides; polyphenols

STUDY DESIGN:
Intervention Model Description: The clinical study will be performed in a double-blind, randomized, monocentric cross-over design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- collagen peptide bovine high molecular weight-Water (Experimental): source: bovine; standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: collagen peptides
- collagen peptide bovine low molecular weight-Water (Experimental): source: bovine; standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: collagen peptides
- collagen peptide bovine low molecular weight- food matrix 1 (Experimental): source: bovine; standardized to 10 g provided as single dose. Orally applied in Food matrix 1
  Interventions: Dietary Supplement: collagen peptides
- collagen peptide bovine low molecular weight- food matrix 2 (Experimental): source: bovine; standardized to 10 g provided as single dose. Orally applied in Food matrix 2
  Interventions: Dietary Supplement: collagen peptides
- collagen peptide fish low molecular weight-Water (Experimental): source: fish; standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: collagen peptides
- collagen peptide porcine low molecular weight-Water (Experimental): source: porcine; standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: collagen peptides

INTERVENTIONS:
Dietary Supplement: collagen peptides — Collagen peptides will be orally administered and pharmacokinetic parameters will be assessed up to 6 hours after study product intake.

SUMMARY:
The aim of this study is the comparison of the oral bioavailability of hydroxyproline, a key marker for collagen peptide intake, after ingestion of collagen peptides from different sources, sizes and together with different food matrices, either containing high or low levels of polyphenols.

DETAILED DESCRIPTION:
The absorption (blood) of collagen peptides from bovine, fish and porcine source in different sizes and administered together with foods of different polyphenol content will be assessed. Pharmacokinetic parameters (AUC0-6h, Cmax and Tmax) after oral single dose administration will be determined to estimate the impact of different sources, different peptide sized any food matrix.

The following objectives will be evaluated exploratory by comparison of pharmacokinetic parameters from the concentration time curve of hydroxyproline, a key marker of collagen type I, between:

* different sources of collagen peptides (bovine, fish, porcine)
* different sizes of collagen peptides from cattle
* food matrices impact on uptake of bovine collagen peptides (dissolved in water vs. food matrix 1 vs. food matrix 2).

Additionally, concentration time curves of further amino acids will be assessed descriptively.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Sex: female and male (50 % of each gender)
* Age: 18-50 years
* BMI ≥19 and ≤28 kg/m²
* Nonsmoker

Main Exclusion Criteria:

* Relevant history or presence of any severe medical disorder, potentially interfering with this study (e.g. mal absorption, chronic gastro-intestinal diseases, heavy depression, diabetes, acute cancers within last 3 years except basal cell carcinoma of the skin, etc.)
* Significant changes in lifestyle or medication (within last 3 mo.) or surgical intervention or surgical procedure such as bariatric surgery
* Application of corticoids (intravenously, orally or intraarticularly) and other immune-suppressing drug (within last 2 weeks)
* Blood donation within 1 month prior to study start or during study
* Regular intake of drugs or supplements possibly interfering with this study (Glucosamine, chondroitin sulfate, hyaluronic acid, omega-3, folic acid, curcumin/turmeric, Boswellia serrata, collagen, Vitamin D) within 2 weeks prior to study start or during study
* Intake of anticoagulants like Heparin, Marcumar etc.
* Coffee consumption >3 cups / day
* History of hypersensitivity to fish

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC(0-6h)) for hydroxyproline after single dose of the different collagen peptides. | pre dose and up to 6 hours post dose
  Pharmakokinetic variable
Peak plasma concentration after administration (Cmax) for hydroxyproline after single dose of the different collagen peptides | pre dose and up to 6 hours post dose
  Pharmakokinetic variable
Time to reach the maximum concentration of hydroxyproline (Tmax) | pre dose and up to 6 hours post dose
  Pharmakokinetic variable

SECONDARY OUTCOMES:
Concentration-time of essential and not essential amino acids | pre dose and up to 6 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No